CLINICAL TRIAL: NCT03350048
Title: Evaluation of Host Biomarker-based Point-of-care Tests for Targeted Screening for Active TB
Acronym: ScreenTB
Status: Completed | Type: Observational
Sponsor: Prof Gerhard Walzl (Other)
Collaborators: Armauer Hansen Research Institute, Ethiopia (Other); Medical Research Council Unit, The Gambia (Other); Leiden University Medical Center (Other); Makerere University (Other); London School of Hygiene and Tropical Medicine (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); LINQ Management GMBH (Unknown)
Responsible Party: Sponsor-Investigator, Prof Gerhard Walzl, Prof, University of Stellenbosch
Organization: University of Stellenbosch (Other)
Other Study IDs: N16/05/070
Record Dates: First submitted 2017-11-17; First posted 2017-11-22 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Pulmonary Tuberculosis
Keywords: Tuberculosis; Point-of-care test; Diagnostics; Biomarkers
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood
  * Sputum
  * Urine
  * Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training Set: First 500 participants recruited for the Training Set:
  * Blood collection for optimization and validation (vs ELISA) of TransDot point-of-care test at LUMC and later for lab-based TransDot at local site laboratory
  * Blood, sputum, saliva and urine collection for secondary objectives and repository
- Test Set: Subsequent 300 participants to be used for the Test Set:
  * Fingerprick TransDot point-of-care test performed at field site after symptom screen and clinical evaluation and before CXR
  * Blood, sputum, saliva and urine collection for secondary objectives and repository
  Interventions: Diagnostic Test: Trans-Dot point-of-care test

INTERVENTIONS:
Diagnostic Test: Trans-Dot point-of-care test — Training set participants will be recruited and receive investigations for TB. Blood samples will also be collected from them for performance of ELISAs and laboratory-based TransDot tests. These blood samples will be drawn at baseline, week 8 and week 24 at end of treatment for confirmed TB cases and at baseline for non-TB cases.
  Test set participants will be recruited and receive investigations for TB. A POC TransDot test will be performed on fingerprick blood at baseline, and at week 8 and week 24 in participants on TB treatment, as well as a laboratory based TransDot test on serum at baseline. The week 8 and week 24 TransDot tests will be used to investigate the test's utility as an indicator of treatment response.
  Groups: Test Set

SUMMARY:
Title: Evaluation of host biomarker-based point-of-care tests for targeted screening for active TB (Screen TB)

Introduction: Tuberculosis (TB) places severe pressure on health care services of the developing world. Despite the introduction of the highly sensitive and specific GeneXpert MTB/RIF (GeneXpert) test [1] with a potential turn-around time of two hours, many people in high TB prevalence areas still do not have access to efficient TB diagnostic services due to logistical constraints in these settings. A cost effective, rapid, point-of-care screening test with high sensitivity would identify people with a high likelihood for active TB and would prioritize them for testing with more expensive, technically or logistically demanding assays including GeneXpert or liquid culture, facilitating cost-effective diagnostic work-up in resource-limited settings. A serum cytokine signature for active TB disease, discovered in the AE-TBC project, with a sensitivity of 89% (CI 78 - 95%) and specificity of 76% (CI 68 - 83%), will be optimised and utilized in a point-of-care format (TransDot) to rapidly test for TB disease in symptomatic people.

Hypothesis: The TransDot test will achieve a sensitivity of > 90% for TB disease, in a training set of people suspected of having TB disease, and be validated (achieve similarly high sensitivity) subsequently in a prospective test set of people suspected of having TB disease, when compared to a composite gold standard of sputum culture, smear, GeneXpert, chest X-ray, TB symptoms and TB treatment response.

Objectives: The overall objective of the study is to incorporate a six-marker serum signature into a multiplex UCP-LFA format, referred to as TransDot, for finger-prick blood testing. The end point of the study is the accuracy (sensitivity and specificity) of the UCP-LFA TransDot test on finger-prick blood for active TB and will be prospectively compared against gold standard composite diagnostic criteria (GeneXpert, MGIT culture, TB sputum smear, CXR, TB symptom screen and response to TB treatment).

Primary: The primary outcome of interest will be accuracy, sensitivity and specificity of the TransDot finger-prick test when compared with the composite gold standard tests.

DETAILED DESCRIPTION:
Protocol Summary Title: Evaluation of host biomarker-based point-of-care tests for targeted screening for active TB (Screen TB)

Population: A total of 800 people presenting at primary health care clinics with presumed active pulmonary tuberculosis, aged 18 to 70 years, male or female gender, will be recruited. They should be willing to give informed, written consent, including consent for HIV testing. They should have symptoms that could be compatible with active TB (cough > two weeks, plus at least one of the following: fever, weight loss, haemoptysis and night sweats). Participants should not have been on TB treatment for the past 90 days and should not have received immune suppressive therapy, be known with alcohol of drug abuse, have a haemoglobin level <9g/dl or be pregnant or breastfeeding. HIV co-infection is not an exclusion criterion. Participants will be recruited from primary health care clinics in Cape Town, South Africa, Windhoek in Namibia, Addis Ababa in Ethiopia, Banjul in The Gambia and Kampala in Uganda.

Number of Sites: Five sites

Study Duration: 3 years

Subject Duration: 18 months for TB cases, 2 months for non-TB cases

Objectives:

The overall objective of the study is to incorporate a six-marker serum signature into a multiplex UCP-LFA format, referred to as TransDot, for finger-prick blood testing. The end point of the study is the accuracy (sensitivity and specificity) of the UCP-LFA TransDot test on finger-prick blood for active TB and will be prospectively compared against gold standard composite diagnostic criteria (GeneXpert, MGIT culture, TB sputum smear, CXR, TB symptom screen and response to TB treatment).

ELIGIBILITY:
Inclusion Criteria:

* Symptoms suggestive of TB disease: cough for more than two weeks with fever, malaise, weight loss, night sweats, haemoptysis, chest pain or loss of appetite.
* Willingness to give consent to take part in the study.
* Willingness to undergo HIV testing or be willing to have their HIV infection status disclosed to the study field workers.
* Eighteen years or older and aged 70 years or younger.

Exclusion Criteria:

* Permanent residence in study area for less than 3 months or with no permanent address.
* Pregnancy or breastfeeding.
* HB<9g/l
* On TB treatment currently or in the last ninety days.
* HIV positive patients currently on INH prophylaxis, or in the last ninety days.
* Known quinolone or aminoglicozide antibiotic use reported in the past 60 days.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult participants with suspected active TB disease will be recruited in South Africa, the Gambia, Uganda, Namibia and Ethiopia. Each site will recruit approximately 160 participants with suspected TB, until the desired overall total of about 800 participants is reached. In South Africa, up to 300 participants will be recruited from primary health care clinics (Adriaanse, Elsiesriver, Uitsig, Ravensmead, Fisantekraal, Durbanville and Dunoon) in Cape Town.
  Patients presenting to the health care facility with symptomatic pulmonary disease and a high likelihood of having tuberculosis will be enrolled and followed up for outcome classification. Participants who had previous TB, extra-pulmonary TB in addition to pulmonary TB, drug resistance detected on GeneXpert or culture or other concomitant diseases, will not be excluded from enrolment. Both HIV positive and HIV negative individuals will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 969 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of the TransDot finger-prick test | 3 years
  The primary outcome of interest will be accuracy, sensitivity and specificity of the TransDot finger-prick test when compared with the composite gold standard tests.

SECONDARY OUTCOMES:
POC TransDOT test versus lab-based tests | 3 years
  To evaluate the agreement between the POC TransDot test and laboratory based ELISAs first (both on serum), and subsequently between POC TransDot (on fingerprick blood) and laboratory based TransDot (on serum).
TransDOT as treatment response marker | 3 years
  To investigate the utility of a TransDot test at month 2 and month 6 as a marker of treatment response.
Identification of additional host marker signatures | 3 years
  To identify additional host marker signatures that can be utilized for future improvement of diagnostic tests in the TransDot format or other point-of care tests that might become available in the future
Evaluation of the serum signature's underlying biological processes | 3 years
  To evaluate the biological processes (cell-based immune profile and components) underlying the six-marker serum signature model during TB disease and treatment response. In parallel, the peripheral profile will compare this to the corresponding profile at the lung infection site.
Optimisation of ultra-sensitive TB culture techniques | 3 years
  To refine and optimise ultra-sensitive TB culture techniques on sputum and compare these to standard techniques and the TransDot test results, at baseline and month 6.
Biomarker Biorepository Samples | 3 years
  To collect appropriate additional host samples for future biomarker research

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Walzl, PhD, MD, Principal Investigator — Head of Department of Biomedical Sciences
Locations (10):
- Armauer Hansen Research Institute, Addis Ababa, Ethiopia
- Germany (2):
  - European Research and Project Office GmbH, Saarbrücken, Saarland
  - LINQ Management GmbH, Berlin
- University of Namibia, Windhoek, Namibia
- Netherlands (2):
  - The European & Developing Countries Clinical Trials Partnership Association (EDCTP), The Hague, South Holland
  - Leiden University Medical Center (Academisch Ziekenhuis Leiden, LUMC), Leiden
- Stellenbosch University, Cape Town, Western Cape, South Africa
- Medical Research Council The Gambia, Banjul, The Gambia
- Makerere University, Kampala, Uganda
- London School of Hygiene and Tropical Medicine, London, United Kingdom

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-05): https://cdn.clinicaltrials.gov/large-docs/48/NCT03350048/Prot_SAP_000.pdf